CLINICAL TRIAL: NCT04169828
Title: The Ondansetron Premedication Trial in Juvenile Idiopathic Arthritis
Acronym: OPT-JIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Arthritis Society, Canada (Other); University of Calgary (Other); The Hospital for Sick Children (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); London Health Sciences Centre (Other); University of Manitoba (Other); Alberta Children's Hospital (Other); McMaster University (Other); McMaster Children's Hospital (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Jaime Guzman, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H18-03176
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Arthritis; Arthritis, Juvenile; Joint Diseases; Rheumatic diseases; Pragmatic Trials; Ondansetron; Methotrexate; Nausea
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis; Joint Diseases; Rheumatic Diseases; Nausea | interventions — Methotrexate; Ondansetron; Leucovorin

STUDY DESIGN:
Intervention Model Description: Pragmatic RCTs use alternative designs to establish effectiveness of a treatment strategy in usual care. Pragmatic trials aim to include all subjects in whom the treatment may be used and are conducted under the usual conditions of practice to demonstrate effectiveness under real word circumstances. Patients enrolled in a pragmatic trial are more representative because eligibility criteria are less strict.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron premedication (Experimental): Methotrexate and folic/folinic acid as prescribed by physician. Ondansetron: 2 mg if <15Kg, 4 mg if 15-30Kg, 8 mg if >30Kg to be taken by mouth one hour before each weekly methotrexate dose, followed by two additional doses every 6-8 hours if awake. To be started from the very first dose of methotrexate.
  Interventions: Drug: Methotrexate; Drug: Ondansetron; Drug: Folic/folinic acid
- Ondansetron as needed (Active Comparator): Methotrexate and folic/folinic acid as prescribed by physician. ONLY children who report nausea/vomiting during regular care will be prescribed ondansetron at the same dose as in experimental group (2 mg if <15Kg, 4 mg if 15-30Kg, 8 mg if >30Kg to be taken by mouth one hour before each weekly methotrexate dose, followed by two additional doses every 6-8 hours if awake), as per the attending rheumatologist's discretion
  Interventions: Drug: Methotrexate; Drug: Ondansetron; Drug: Folic/folinic acid

INTERVENTIONS:
Drug: Methotrexate — Children in both the intervention and control group will receive Methotrexate dosed as prescribed by the attending rheumatologist
  Other Names: Trexall
Drug: Ondansetron — Children in the intervention group will be prescribed premedication with oral ondansetron.
  Children in the control group will be prescribed ondansetron ONLY if the child reports nausea/vomiting during regular treatment care with Methotrexate
  Other Names: Zofran
Drug: Folic/folinic acid — Children in both intervention and control group will receive folic acid or folinic acid dosed as prescribed by the attending rheumatologist.
  Other Names: Leucovorin

SUMMARY:
Far too many kids and families live in dread over the weekly nausea and vomiting caused by methotrexate - a medicine that controls joint swelling in Juvenile Arthritis patients. If methotrexate is not tolerated, expensive alternative biological medications may be started. This registry-based pragmatic randomized controlled trial will evaluate if routine premedication with the anti-emetic drug Ondansetron, reduces nausea and vomiting and increases the proportion of children able to continue methotrexate. By preventing nausea before it starts, the investigators hope to give kids and families a better quality of life and see a more cost-effective use of medication.

DETAILED DESCRIPTION:
1. Purpose:

   To evaluate if routine pre-medication with the anti-emetic ondansetron reduces methotrexate intolerance and increases the proportion of children with JIA able to continue taking methotrexate, resulting in a better quality of life and more cost-effective medication use.
2. Hypothesis:

   Prophylactic prescription of ondansetron with methotrexate will increase the proportion of children that remain on methotrexate and intolerance free one year after starting methotrexate, relative to prescription of ondansetron after intolerance symptoms develop.
3. Justification:

   Methotrexate intolerance is thought to be largely the result of Pavlovian conditioning secondary to previous exposure and symptoms can be triggered by associated stimuli, such as a yellow liquid similar in color to methotrexate or the smell of alcohol cleansing swabs. This intolerance leads to poor adherence to optimal dosing or to stopping the medication altogether. Children who cannot adhere to optimal dosing or stop methotrexate may require expensive biologic medications to control their JIA. Methotrexate intolerance often leads to use of anti-emetic medications which, unfortunately, rarely reverse conditioned responses. In oncology anti-emetics are used prophylactically as premedication in all subjects receiving chemotherapy to prevent the establishment of conditioned intolerance.

   By conducting a registry-based pragmatic adaptive superiority randomized clinical trial the investigators will include most subjects in whom the treatment may be used under the usual conditions of practice to demonstrate effectiveness under real word circumstances. Patients enrolled in a pragmatic trial are more representative because eligibility criteria are less strict. More so, a registry-based pragmatic RCT can also be much cheaper than a traditional RCT.
4. Objectives:

The investigators will assign patients starting low-dose methotrexate for JIA 1:1 online using the CAPRI Registry and block randomization by Canadian region and patient weight to one of two groups:

Intervention: Routine premedication with oral ondansetron (2, 4 or 8 mg for patient weights <15Kg, 15-30Kg, >30 Kg; 3 doses a week).

Control: Oral ondansetron at the same dosing, prescribed only to those patients who develop methotrexate-induced nausea/vomiting during usual care.

The investigators will compare:

1. The proportions of patients remaining on methotrexate with no intolerance between the two groups one year after starting methotrexate (primary objective).
2. Safety and tolerability
3. The cumulative incidence of:

   1. methotrexate intolerance
   2. attainment of inactive disease
   3. biologic medication initiation
4. The mean quality of life scores and methotrexate intolerance severity scores between the two groups 4-8 months after starting methotrexate.

   The investigators will also collect information on impacts on quality of life and medication utilization that will enable a future cost-effectiveness analysis.
5. Research Design:

   The investigators will conduct a CAPRI JIA Registry-based pragmatic adaptive superiority RCT as per the following methods.

   Registry-based: The trial will use infrastructure already in place for the CAPRI JIA Registry.

   Pragmatic: Broad inclusion criteria and simple outcome assessments compatible with usual care.

   Adaptive: This is a Planned Sample-Size Re-Estimation Adaptive Trial as described by Bhatt & Metha [34].

   Superiority: Designed to test superiority (as opposed to non-inferiority) of ondansetron premedication.

   RCT: Treatments assigned by block randomization and analyses adjusted for post-randomization imbalances
6. Statistical Analysis:

The primary outcome statistic is the ratio of two proportions (relative risk, RR), the proportion of children remaining on methotrexate with no intolerance in the intervention group divided by the same in the control group. This choice allows flexibility for the frequency of follow-up visits to be set-up as per clinical need, obviating the need for study-specific visits, increasing feasibility and decreasing costs. It is also not impacted by the times at which methotrexate intolerance or discontinuation occur which leads to simplicity in interpretation and analysis.

The sample size calculation is based on expressing the RR in the log scale and using established formulas for standard errors. With p<0.05, power of 90% and expected methotrexate continuation with no intolerance of 50% in the control group and 75% in the intervention group the result is 79 evaluable subjects per group. The investigators will aim to recruit 176 subjects total to allow for up to a 10% dropout rate, although they expect a dropout rate of <5% based on previous CAPRI studies.

A preliminary analysis after recruitment of 90 subjects will consist of a two-sided confidence interval (CI) for the RR of continuing on methotrexate with no intolerance, where the confidence level is adjusted for information accrual as per Schoenfeld.

The Data and Safety Committee will assess preliminary results according to the following guidance:

If the CI is entirely below a relative risk of 1.2, the study will be stopped for futility.

If the CI is entirely above a relative risk of 1.2, the study will be stopped and superiority will be claimed.

If the CI includes a relative risk of 1.2, the trial will continue until the re-calculated full target sample is attained.

The RR of 1.2 has been selected on clinical grounds. In a prospective study of 142 children with JIA starting methotrexate followed for one year, Van Dijkhuizen et al reported that 59 patients developed intolerance and 11 discontinued methotrexate for other reasons, for a total of 72 (50.7%) remaining on methotrexate with no intolerance. An increase in this proportion to <60% is deemed too small to justify the additional costs and risks of adding prophylactic ondansetron.

The final analysis will be an intention to treat analysis conducted after the final sample size is achieved or at the time the study is stopped. All subjects enrolled in the study at that time will complete a one-year follow-up and will be included in the final analysis. Logistic regression models will be used to adjust effect estimates for post-randomization imbalances in the two groups (intervention, control). A secondary per-protocol analysis will be conducted on those subjects who received the assigned intervention for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 4-16 years
2. Diagnosis of JIA as per ILAR criteria [1], irrespective of JIA category
3. Followed at a CAPRI centre in Canada
4. Starting methotrexate to control JIA manifestations (arthritis, uveitis, psoriasis). (Female subjects of child bearing potential who are taking methotrexate for JIA cannot be pregnant, breastfeeding, or planning a pregnancy while on the drug and females of childbearing potential who are sexually active must use highly effective medically acceptable contraception. Subjects who stop methotrexate during the study will also discontinue ondansetron.)
5. Informed written consent to participate
6. Participating in the CAPRI JIA Registry

Exclusion Criteria:

1. Previous use of methotrexate
2. Known hypersensitivity to ondansetron or any components of its formulations
3. Known hypersensitivity to other 5-HT3 antagonists
4. Known congenital Long-QT syndrome
5. Patients taking other medicinal products that lead to either QT prolongation or electrolyte abnormalities
6. Because the serotonin syndrome may occur when ondansetron is combined with other agents that may affect the serotonergic neurotransmitter system, patients receiving any of the serotonergic and/or neuroleptic drugs listed below will be excluded:

   • Triptans, SSRIs, SNRIs, lithium, sibutramine, fentanyl and its analogues, dextromethorphan, tramadol, tapendalol, meperidine, methadone, pentazocine or St. John's Wort (Hypericum perforatum), MAOIs, linezolid, methylene blue.
7. Patients who are pregnant or breastfeeding, or are sexually active and unwilling to practice an acceptable method of birth control.
8. Family unable to complete questionnaires in English or French

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that remain on methotrexate with no intolerance | One year after starting methotrexate.
  Intolerance will be defined as ≥6 points in the English or French versions of the validated Methotrexate Intolerance Severity Score, MISS [10, 36]. Scores in the MISS questionaire go from 0 (no signs of intolerance) to a maximum of 36 (all signs of intolerance are severe). The MISS questionnaire takes less than 2 minutes to complete (see Appendix). It will be added to the Registry questionnaires completed by families online or on paper as per the CAPRI Centre usual Registry procedures.

SECONDARY OUTCOMES:
Frequency and cumulative incidence of adverse events (safety and tolerability) | Within one year
  Frequency and cumulative incidence of adverse events, and any suspected unexpected serious adverse drug reactions (SUSARs).
Methotrexate intolerance | Within one year
  The cumulative incidence of methotrexate intolerance
Attainment of inactive disease | Within one year
  The cumulative incidence of attainment of inactive disease, defined by Wallace criteria
Starting a biologic medication | Within one year
  The cumulative incidence of starting a biologic medication
Quality of My Life scale | 4-8 months after starting methotrexate
  Mean quality of life scores in the Quality of My Life scale. The scale has a minimum value of zero (WORST quality of life) and a maximum value of 10 (BEST quality of life).
MISS questionnaire | 4-8 months after starting methotrexate
  Mean scores in the Methotrexate Intolerance Severity Score (MISS) questionnaire. Scores in the MISS questionnaire go from 0 (no signs of intolerance) to a maximum of 36 (all signs of intolerance are severe).

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Guzman, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (11):
- Canada (11):
  - University of Calgary / Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - University of Manitoba/Children's hospital research institute, Winnipeg, Manitoba
  - McMaster University/McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Université de Montréal, Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
If the ethics boards at all participating centres approve individual participant data sharing we will upload to clinicaltrials.gob a data sharing plan at that time.

REFERENCES:
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] Shiff NJ, Lix LM, Joseph L, Duffy C, Tucker LB, Svenson LW, Belisle P, Bernatsky S. The prevalence of systemic autoimmune rheumatic diseases in Canadian pediatric populations: administrative database estimates. Rheumatol Int. 2015 Mar;35(3):569-73. doi: 10.1007/s00296-014-3136-6. Epub 2014 Sep 26. PMID 25257764
- [Background] ANSELL BM, BYWATERS EG. RHEUMATOID ARTHRITIS (STILL'S DISEASE). Pediatr Clin North Am. 1963 Nov;10:921-39. doi: 10.1016/s0031-3955(16)31475-4. No abstract available. PMID 14145024
- [Background] Giannini EH, Brewer EJ, Kuzmina N, Shaikov A, Maximov A, Vorontsov I, Fink CW, Newman AJ, Cassidy JT, Zemel LS. Methotrexate in resistant juvenile rheumatoid arthritis. Results of the U.S.A.-U.S.S.R. double-blind, placebo-controlled trial. The Pediatric Rheumatology Collaborative Study Group and The Cooperative Children's Study Group. N Engl J Med. 1992 Apr 16;326(16):1043-9. doi: 10.1056/NEJM199204163261602. PMID 1549149
- [Background] Beukelman T, Patkar NM, Saag KG, Tolleson-Rinehart S, Cron RQ, DeWitt EM, Ilowite NT, Kimura Y, Laxer RM, Lovell DJ, Martini A, Rabinovich CE, Ruperto N. 2011 American College of Rheumatology recommendations for the treatment of juvenile idiopathic arthritis: initiation and safety monitoring of therapeutic agents for the treatment of arthritis and systemic features. Arthritis Care Res (Hoboken). 2011 Apr;63(4):465-82. doi: 10.1002/acr.20460. PMID 21452260
- [Background] Guzman J, Oen K, Tucker LB, Huber AM, Shiff N, Boire G, Scuccimarri R, Berard R, Tse SM, Morishita K, Stringer E, Johnson N, Levy DM, Duffy KW, Cabral DA, Rosenberg AM, Larche M, Dancey P, Petty RE, Laxer RM, Silverman E, Miettunen P, Chetaille AL, Haddad E, Houghton K, Spiegel L, Turvey SE, Schmeling H, Lang B, Ellsworth J, Ramsey S, Bruns A, Campillo S, Benseler S, Chedeville G, Schneider R, Yeung R, Duffy CM; ReACCh-Out investigators. The outcomes of juvenile idiopathic arthritis in children managed with contemporary treatments: results from the ReACCh-Out cohort. Ann Rheum Dis. 2015 Oct;74(10):1854-60. doi: 10.1136/annrheumdis-2014-205372. Epub 2014 May 19. PMID 24842571
- [Background] Falvey S, Shipman L, Ilowite N, Beukelman T. Methotrexate-induced nausea in the treatment of juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2017 Jun 19;15(1):52. doi: 10.1186/s12969-017-0180-2. PMID 28629458
- [Background] Bulatovic M, Heijstek MW, Verkaaik M, van Dijkhuizen EH, Armbrust W, Hoppenreijs EP, Kamphuis S, Kuis W, Egberts TC, Sinnema G, Rademaker CM, Wulffraat NM. High prevalence of methotrexate intolerance in juvenile idiopathic arthritis: development and validation of a methotrexate intolerance severity score. Arthritis Rheum. 2011 Jul;63(7):2007-13. doi: 10.1002/art.30367. PMID 21437879
- [Background] Dupont-Lucas C, Grandjean-Blanchet C, Leduc B, Tripcovici M, Larocque C, Gervais F, Jantchou P, Amre D, Deslandres C. Prevalence and Risk Factors for Symptoms of Methotrexate Intolerance in Pediatric Inflammatory Bowel Disease. Inflamm Bowel Dis. 2017 Feb;23(2):298-303. doi: 10.1097/MIB.0000000000001014. PMID 28107279
- [Background] Mulligan K, Wedderburn LR, Newman S. The experience of taking methotrexate for juvenile idiopathic arthritis: results of a cross-sectional survey with children and young people. Pediatr Rheumatol Online J. 2015 Dec 12;13:58. doi: 10.1186/s12969-015-0052-6. PMID 26653415
- [Background] van Dijkhuizen EH, Bulatovic Calasan M, Pluijm SM, de Rotte MC, Vastert SJ, Kamphuis S, de Jonge R, Wulffraat NM. Prediction of methotrexate intolerance in juvenile idiopathic arthritis: a prospective, observational cohort study. Pediatr Rheumatol Online J. 2015 Feb 18;13:5. doi: 10.1186/s12969-015-0002-3. eCollection 2015. PMID 25745368
- [Background] Bechard MA, Lemieux JR, Roth J, Watanabe Duffy K, Duffy CM, Aglipay MO, Jurencak R. Procedural pain and patient-reported side effects with weekly injections of subcutaneous methotrexate in children with rheumatic disorders. Pediatr Rheumatol Online J. 2014 Dec 19;12:54. doi: 10.1186/1546-0096-12-54. eCollection 2014. PMID 25584042
- [Background] Klotsche J, Minden K, Niewerth M, Horneff G. Time spent in inactive disease before MTX withdrawal is relevant with regard to the flare risk in patients with JIA. Ann Rheum Dis. 2018 Jul;77(7):996-1002. doi: 10.1136/annrheumdis-2017-211968. Epub 2018 Feb 16. PMID 29453217
- [Background] Scheuern A, Tyrrell PN, Haas JP, Hugle B. Countermeasures against methotrexate intolerance in juvenile idiopathic arthritis instituted by parents show no effect. Rheumatology (Oxford). 2017 Jun 1;56(6):901-906. doi: 10.1093/rheumatology/kew507. PMID 28122960
- [Background] Schoemaker CG, van Dijkhuizen EHP, Vastert SJ. Contradictory and weak evidence on the effectiveness of anti-emetics for MTX-intolerance in JIA-patients. Pediatr Rheumatol Online J. 2018 Feb 15;16(1):13. doi: 10.1186/s12969-018-0229-x. No abstract available. PMID 29448947
- [Background] Phillips RS, Friend AJ, Gibson F, Houghton E, Gopaul S, Craig JV, Pizer B. Antiemetic medication for prevention and treatment of chemotherapy-induced nausea and vomiting in childhood. Cochrane Database Syst Rev. 2016 Feb 2;2(2):CD007786. doi: 10.1002/14651858.CD007786.pub3. PMID 26836199
- [Background] Cubeddu LX, Hoffmann IS, Fuenmayor NT, Finn AL. Efficacy of ondansetron (GR 38032F) and the role of serotonin in cisplatin-induced nausea and vomiting. N Engl J Med. 1990 Mar 22;322(12):810-6. doi: 10.1056/NEJM199003223221204. PMID 1689807
- [Background] De Mulder PH, Seynaeve C, Vermorken JB, van Liessum PA, Mols-Jevdevic S, Allman EL, Beranek P, Verweij J. Ondansetron compared with high-dose metoclopramide in prophylaxis of acute and delayed cisplatin-induced nausea and vomiting. A multicenter, randomized, double-blind, crossover study. Ann Intern Med. 1990 Dec 1;113(11):834-40. doi: 10.7326/0003-4819-113-11-834. PMID 2146911
- [Background] Dick GS, Meller ST, Pinkerton CR. Randomised comparison of ondansetron and metoclopramide plus dexamethasone for chemotherapy induced emesis. Arch Dis Child. 1995 Sep;73(3):243-5. doi: 10.1136/adc.73.3.243. PMID 7492164
- [Background] Kempinska A, Benchimol EI, Mack A, Barkey J, Boland M, Mack DR. Short-course ondansetron for the prevention of methotrexate-induced nausea in children with Crohn disease. J Pediatr Gastroenterol Nutr. 2011 Oct;53(4):389-93. doi: 10.1097/MPG.0b013e31822855e7. PMID 21681112
- [Background] Blanco R, Gonzalez-Gay MA, Garcia-Porrua C, Ibanez D, Garcia-Pais MJ, Sanchez-Andrade A, Vazquez-Caruncho M. Ondansetron prevents refractory and severe methotrexate-induced nausea in rheumatoid arthritis. Br J Rheumatol. 1998 May;37(5):590-2. doi: 10.1093/rheumatology/37.5.590. No abstract available. PMID 9651100
- [Background] Cubeddu LX, Pendergrass K, Ryan T, York M, Burton G, Meshad M, Galvin D, Ciociola AA. Efficacy of oral ondansetron, a selective antagonist of 5-HT3 receptors, in the treatment of nausea and vomiting associated with cyclophosphamide-based chemotherapies. Ondansetron Study Group. Am J Clin Oncol. 1994 Apr;17(2):137-46. doi: 10.1097/00000421-199404000-00010. PMID 8141105
- [Background] Silverman E, Mouy R, Spiegel L, Jung LK, Saurenmann RK, Lahdenne P, Horneff G, Calvo I, Szer IS, Simpson K, Stewart JA, Strand V; Leflunomide in Juvenile Rheumatoid Arthritis (JRA) Investigator Group. Leflunomide or methotrexate for juvenile rheumatoid arthritis. N Engl J Med. 2005 Apr 21;352(16):1655-66. doi: 10.1056/NEJMoa041810. PMID 15843668
- [Background] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Bhatt DL, Mehta C. Adaptive Designs for Clinical Trials. N Engl J Med. 2016 Jul 7;375(1):65-74. doi: 10.1056/NEJMra1510061. No abstract available. PMID 27406349
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Chausset A, Fargeix T, Pereira B, Echaubard S, Duquesne A, Desjonqueres M, Freychet C, Belot A, Merlin E. MISS questionnaire in French version: a good tool for children and parents to assess methotrexate intolerance. Clin Rheumatol. 2017 Jun;36(6):1281-1288. doi: 10.1007/s10067-017-3638-1. Epub 2017 May 5. PMID 28477218
- [Background] Wallace CA, Giannini EH, Huang B, Itert L, Ruperto N; Childhood Arthritis Rheumatology Research Alliance; Pediatric Rheumatology Collaborative Study Group; Paediatric Rheumatology International Trials Organisation. American College of Rheumatology provisional criteria for defining clinical inactive disease in select categories of juvenile idiopathic arthritis. Arthritis Care Res (Hoboken). 2011 Jul;63(7):929-36. doi: 10.1002/acr.20497. PMID 21717596
- [Background] Feldman BM, Grundland B, McCullough L, Wright V. Distinction of quality of life, health related quality of life, and health status in children referred for rheumatologic care. J Rheumatol. 2000 Jan;27(1):226-33. PMID 10648043
- [Background] Otto C, Barthel D, Klasen F, Nolte S, Rose M, Meyrose AK, Klein M, Thyen U, Ravens-Sieberer U. Predictors of self-reported health-related quality of life according to the EQ-5D-Y in chronically ill children and adolescents with asthma, diabetes, and juvenile arthritis: longitudinal results. Qual Life Res. 2018 Apr;27(4):879-890. doi: 10.1007/s11136-017-1753-8. Epub 2017 Nov 30. PMID 29189988
- [Background] Schoenfeld DA. A simple algorithm for designing group sequential clinical trials. Biometrics. 2001 Sep;57(3):972-4. doi: 10.1111/j.0006-341x.2001.00972.x. PMID 11550952
- See also: Health Canada prescribing information for methotrexate. — https://pdf.hres.ca/dpd_pm/00053618.PDF
- See also: Hopper C, Khan S, Mancini J, Rennick J. Perceptions of Methotrexate Intolerance in School-aged Children With Juvenile Idiopathic Arthritis [abstract].Arthritis Rheumatol. 2017; 69 (suppl 4). — http://acrabstracts.org/abstract/perceptions-of-methotrexate-intolerance-in-school-aged-children-with-juvenile-idiopathic-arthritis/.
- See also: Da Silva C, Farias A, Sinicato N, Veloso R, Marini R, Appenseller S. Reasons for stopping methotrexate treatment in patients with juvenile idiopathic arthritisPediatric Rheumatology 2014, 12(Suppl 1):P199 (abstract) — http://www.ped-rheum.com/content/12/S1/P199
- See also: Health Canada prescribing information for ondansetron — https://pdf.hres.ca/dpd_pm/00058412.PDF
- See also: Ontario Drug Benefit Formulary — https://www.formulary.health.gov.on.ca/formulary/

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT04169828/SAP_000.pdf